CLINICAL TRIAL: NCT00001194
Title: NMR Scanning on Patients
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 840058; 84-CC-0058
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-03

CONDITIONS: Diagnostic Imaging
Keywords: Helium Cryogen; Magnetic Field; Multi-Institute; Nitrogen Cryogen; Radiofrequency

SUMMARY:
This protocol is designed to investigate the use of novel techniques in MRI that may not yet be commercially available. Specifically, the protocol enables patients to take advantage of new pulse sequence software, coil design or post processing capabilities not otherwise available. The informed consent explains MRI in lay terms, describes the use of contrast agents and lists contraindications to MRI.

DETAILED DESCRIPTION:
NMR imaging promises to provide useful and unique diagnostic information in a variety of diseases. In an attempt to evaluate its role, we plan to study a wide range of diseases during the initial year of imaging. Exposure to magnetic fields and radiofrequency energies of this magnitude have demonstrated no deleterious effects clinically or in the laboratory. The only restrictions will be those imposed by ferromagnetic objects within the patient which would increase the risk of placing them in a strong magnetic field.

ELIGIBILITY:
Any patient undergoing MRI for research or clinical purposes who is participating in a currently active NIH protocol.

No patients with pacemakers, cochlear implants, implanted pumps, shrapnel, metal in the globe of the eye, cerebral aneurysm clips or other contraindication to MRI.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99999
Dates: Start 1984-04; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Choyke PL, Walther MM, Wagner JR, Rayford W, Lyne JC, Linehan WM. Renal cancer: preoperative evaluation with dual-phase three-dimensional MR angiography. Radiology. 1997 Dec;205(3):767-71. doi: 10.1148/radiology.205.3.9393533.
- [Background] Niendorf HP, Dinger JC, Haustein J, Cornelius I, Alhassan A, Clauss W. Tolerance data of Gd-DTPA: a review. Eur J Radiol. 1991 Jul-Aug;13(1):15-20. doi: 10.1016/0720-048x(91)90049-2. PMID 1889423